CLINICAL TRIAL: NCT02956317
Title: A Randomized, Double-Blind, Within-Subject Placebo Controlled Study to Evaluate the Safety and Efficacy of Various Doses of STP705 Administered as Intradermal Injection in Subjects With Hypertrophic Scar.
Brief Title: A Randomized Study to Evaluate the Safety and Efficacy of Various Doses of STP705 in Subjects With Hypertrophic Scar
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SRN-705-001
Record Dates: First submitted 2016-10-31; First posted 2016-11-07 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2017-11

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- STP705 (Active Comparator): Each subject will receive both active (STP705) and control (Placebo) intradermal injection twice a week for a total of 4 weeks at 20 μg/cm2/day (in Cohort A), 30 μg/cm2/day (in Cohort B) and 40 μg/cm2/day (in cohort C). The total length of linear hypertrophic scar will be divided equally for treatment with STP705 and placebo. STP705 and Placebo will be injected intradermal every 1 cm length on the hypertrophic scar.
  Interventions: Drug: STP705; Drug: Placebo
- Placebo (Placebo Comparator): Each subject will receive both active (STP705) and control (Placebo) intradermal injection twice a week for a total of 4 weeks at 20 μg/cm2/day (in Cohort A), 30 μg/cm2/day (in Cohort B) and 40 μg/cm2/day (in cohort C). The total length of linear hypertrophic scar will be divided equally for treatment with STP705 and placebo. STP705 and Placebo will be injected intradermal every 1 cm length on the hypertrophic scar
  Interventions: Drug: STP705; Drug: Placebo

INTERVENTIONS:
Drug: STP705 — The Cotsiranib drug substance is composed of two siRNA oligonucleotides, targeting TGF-β1 and Cox-2 mRNA respectively, and formulated in nanoparticles with Histidine-Lysine co-Polymer (HKP) peptide at a ratio of 1:4 in mass weight (siRNA:peptide), which is further formulated into a dry powder drug product. The administration route would be intra-dermal injection.
  Other Names: COTSIRANIB
Drug: Placebo — Normal Saline

SUMMARY:
This is a randomized, double-blind, within-subject placebo controlled study to evaluate the safety and efficacy of various doses of STP705 administered as intradermal Injection in subjects with hypertrophic scar. The goals are to determine the recommended Phase 2 dose, the pharmacokinetics and pharmacidynamics parameters, and conduct analysis of biomarkers common to the scar formation pathway.

DETAILED DESCRIPTION:
This single-center, randomized, double-blind, within-subject placebo controlled study is designed to evaluate the safety and efficacy of various doses of STP705 administered as intradermal injection in subjects with linear hypertrophic scar.

Twenty four subjects will be divided equally among 3 cohorts (20, 30 and 40 μg/cm2/day dose level) of 8 subjects each. Each subject will receive both active (STP705) and control (Placebo) treatment twice a week for a total of 4 weeks. The total length of linear hypertrophic scar will be divided equally for treatment with STP705 and placebo. STP705 and Placebo will be injected intradermal every 1 cm length on the hypertrophic scar.

Subjects will be confined to clinic or research unit for 24 hours post-dosing after the first treatment administration for the serial PK assay and the blood sample will be collected at the following post-dosing times: 30 min, 1 hr, 2 hrs, 3 hrs, 4 hrs, 5hrs, 6 hrs, 8 hrs, 12 hrs, 16 hrs, 24 hrs, 32 hrs and 36 hrs. Post-dosing ECG will be performed 6 hours (±1 hr) after the first study drug administration and vital signs will be monitored every 2h till 12h post-administration. Adverse events and medications will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to understand and willing to conform to the study procedures and has signed the informed consent form (ICF).
2. Subject is male or female, between the ages of 18 and 60 years, inclusive.
3. Subject with a hypertrophic scar that meet all of the following criteria:

   * linear scar, ≥5 to ≤40 cm in length (Cohort A), ≥5 to ≤50 cm in length (Cohort B), ≥5 to ≤60 cm in length (Cohort C)
   * present for minimum 6 months and no greater than 24 months
   * located anywhere in the body except on the face or front of neck
   * resulting from surgical or traumatic injury
4. Subject is judged, by the Investigator, to be healthy as evidenced by lack of clinically significant abnormal findings on medical history, physical examination, electrocardiogram, vital signs, and clinical laboratory tests.
5. Subject is willing and able to complete the entire course of the trial and to comply with the trial instructions.
6. Subject, if female of child-bearing potential, has a negative serum pregnancy test at screening and a negative urine pregnancy test at prior to treatment and willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence) throughout the study.

Exclusion Criteria:

1. Subjects identified as having keloid or burn scars
2. Subjects who are positive for hepatitis B surface antigen (HbsAg), hepatitis C antibody and HIV.
3. Concurrent use of corticosteroids (including inhaled steroids) and COX-2 inhibitors
4. Are immuno-compromised (HIV infected, cancer and other disease affecting the basal immune response)
5. Clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, hematological, or metabolic disease that is, in the opinion of the Investigator, not stabilized or may otherwise impact the results of the study.
6. Known allergy or hypersensitivity to the study drug(s) or one of the ingredients of the formulation.
7. Any infection or wound in the area to treat.
8. Female subjects who are pregnant or breast-feeding.
9. Participation in a clinical study involving administration of an investigational compound within the past 30 days.
10. Existence of any surgical, medical or laboratory condition that, in the judgment of the clinical investigator, might interfere with the safety, distribution, metabolism or excretion of the drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Differences among the 3 dosage Groups in 24 Patients' appearance of the scar from baseline evaluated by Patient and Observer Scar Assessment Scale (POSAS) | 32 weeks

SECONDARY OUTCOMES:
Change in appearance of the scar from baseline evaluated by Physician Global Assessment using Physician Overall Opinion Question of Patient and Observer Scar Assessment Scale (POSAS) at T4, T8, FU1, FU2 and FU3 visits. | 32 weeks
  Physician global assessment will be performed using the overall opinion question of the POSAS scale. Physicians will be asked to rate the severity of the participant's scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (worst imaginable scar). Within participant treatment difference from baseline will be assessed separately for Site A and Site B.
Change in appearance of the scar from baseline evaluated by Physician Scar Assessment using Complete Patient and Observer Scar Assessment Scale (POSAS) at T4, T8, FU1, FU2 and FU3 visits. | 32 weeks
  Within participant treatment difference from baseline will be assessed separately for Site A and Site B.
Change in appearance of the scar from baseline evaluated by Patient Global Assessment Using Overall Opinion of Patient and Observer Scar Assessment Scale (POSAS) at T4, T8, FU1, FU2 and FU3 visits | 32 weeks
  Patient global assessment was performed using the overall opinion question of the POSAS scale.
  Participants were asked to rate the severity of their scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (very different from normal skin). Within participant treatment difference from baseline will be assessed separately for Site A and Site B.
Change in volume/size of the scar from baseline evaluated by volumetric measurement using 3D camera at T4, T8, FU1, FU2 and FU3 visits | 32 weeks
  Within participant treatment difference from baseline will be assessed separately for Site A and Site B.

OTHER OUTCOMES:
Safety and Tolerability as measured by adverse events (AEs) and clinically relevant changes in laboratory values, vital signs, electrocardiograms (ECGs), and physical examination variables | 32 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided